# Amplifying Consequences to Reduce Dietary Restriction: A Proof-of-Concept Study

NCT06598111

12/14/2023

**Title of research study:** Imagining the Future

Investigator: Lauren M. Harris

Faculty Advisor: Thomas Joiner

**<u>Key Information</u>**: The following is a short summary of this study to help you decide whether or not to be a part of this study. More detailed information is listed later on in this form.

### Why am I being invited to take part in a research study?

We invite you to take part in a research study because you volunteered as a potential participant. You are eligible for this study because you indicated concerns related to your eating or weight.

### What should I know about a research study?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

### Why is this research being done?

The purpose of this study is to evaluate the effects of thinking about the future on behaviors in the short-term.

### How long will the research last and what will I need to do?

We expect that you will be in this research study for 7 days.

The entire study will take place online. You will be asked to (a) read and sign a consent form if you agree to participate; (b) complete a few brief questionnaires; (c) complete a task that involves imagining a day in the future, then writing and reading aloud a short description of this future day; (c) repeat these procedures every 24 hours until you have participated for a total of 7 days; and (d) you will be debriefed and compensated with research study credit.

More detailed information about the study procedures can be found under "What happens if I say yes, I want to be in this research?"

### Is there any way being in this study could be bad for me?

This study has the risk of causing distress while completing questionnaires or reading and writing about sensitive topics. We do not expect any discomfort to last more than a few minutes. There is also a very minimal risk of breach of confidentiality during this study. The researchers have taken several steps to minimize potential risks. You are free to contact the principal investigator by email to discuss any emotional distress that you may experience during participation.

More detailed information about the risks of this study can be found under "Is there any way being in this study could be bad for me? (Detailed Risks)"

### Will being in this study help me in any way?

We cannot promise any benefits to you or others from your taking part in this research, other than compensation. However, it is possible that your participation may serve to help others in the future.

### What happens if I do not want to be in this research?

Participation in research is completely voluntary. You can decide to participate or not to participate.

Earning course or other academic credit by taking part in this study may be an alternative to the requirement that you otherwise complete a course, paper or other credit-earning activity.

Instead of being in this research study, your choices may include: participating in a different research study, or opting not to participate in research. Other studies may have their own unique risks and benefits.

**<u>Detailed Information:</u>** The following is more detailed information about this study in addition to the information listed above.

#### Who can I talk to?

If you have questions, concerns, or complaints, or think the research has hurt you, you may talk to the research team. The researcher conducting this study is Lauren M. Harris, M.S. in the Department of Psychology in Florida State University. If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team at <a href="mailto:harris@psy.fsu.edu">harris@psy.fsu.edu</a>.

This research has been reviewed and approved by an Institutional Review Board ("IRB"). You may talk to them at 850-644-7900 or humansubjects@fsu.edu if:

- Your questions, concerns, or complaints are not being answered by the research team.
  - You cannot reach the research team.
  - You want to talk to someone besides the research team.
  - You have questions about your rights as a research subject.
  - You want to get information or provide input about this research.

## How many people will be studied?

We expect about 200 people will be included in this research study.

## What happens if I say "yes" to being in this research?

- 1) All study procedures will take place online. Before beginning the study, you will be asked to review and sign a consent form received electronically.
- 2) After providing informed consent, you will be asked to complete a series of questionnaires via online survey software. In addition to these questionnaires, you may be asked to read a written excerpt and answer a series of True or False comprehension questions about what you read.
- 3) Next, you will be asked to vividly imagine a hypothetical future scenario and write a verbal description (~300 words) of what you imagined. You will also be asked to provide a voice recording of you reading your response aloud.
- 4) You will complete questionnaires and submit voice recordings each day for a total of 7 days. You will receive a link to participate each day and will have a 24-hour window during which to complete study procedures after you receive the link.
- 5) Upon completion of study procedures, you will be debriefed, provided with mental health resources, and compensated with SONA credit.

The specific tasks you complete will vary slightly depending on your study condition, which will be chosen by chance, like flipping a coin. Neither you nor the researchers will choose which condition you are placed in. You will have an equal chance of being placed in each condition. You will not be told which condition you are placed in; however, the research team will know.

Please note that you may not be made aware of some features about the study, such as its exact purpose, study questions and materials, or your responses that we would like to collect. At the end of your participation in this study or if you withdraw from this study we will provide you with additional information.

### What are my responsibilities if I take part in this research?

If you take part in this research, you will be responsible for completing daily online surveys. This will require you to check your email regularly. You must have consistent internet access to participate in this online study, as well as access to a computer or smartphone with a microphone and audio recording capabilities.

## What happens if I say "yes," but I change my mind later?

You can leave the research at any time it will not be held against you.

### Is there any way being in this study could be bad for me? (Detailed Risks)

There is a risk that you might feel upset when responding to some of the questionnaire items or while completing study tasks. There is also a very minimal risk of breach of confidentiality during this study.

Neither you nor your insurance company will be charged for the services performed in this research study.

## What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study and medical records, to people who have a need to review this information. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB and other representatives of this organization. Your information collected as a part of this research study will not be used or distributed for future research studies.

We may publish the results of this research. However, we will keep your name and other identifying information confidential to the extent allowed by law.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### What else do I need to know?

If you agree to take part in this online research study, you will be provided with SONA credit for your time and effort. You will receive 1 SONA credit for completing the first survey and follow-up, and an additional 0.5 SONA credits for each subsequent day you participate in the study, for a total of 3.5 SONA credits. You may receive an additional 0.5 "bonus" SONA credit if you complete all 7 days of the study and follow all study instructions correctly, for a total of 4 SONA credits.

Instead of being in this research study, your choices may include: participating in a different research study, or opting not to participate in research. Other studies may have their own unique risks and benefits.

## **Signature Block for Capable Adult**

Your signature documents your permission to take part in this research.

Signature of subject

Date

Printed name of subject

Signature of person obtaining consent

Date